CLINICAL TRIAL: NCT00741117
Title: The Influence of Conjugated Hyperbilirubinemia on Pulse Oximetric Accuracy in Liver Disease
Brief Title: Conjugated Hyperbilirubinemia and Pulse Oximetry
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to insufficient personnel required to conduct trial.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ram Subramanian, M.D. Department of Medicine, Hepatology, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00008493
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Liver Disease; Hyperbilirubinemia
Keywords: Pulse Oximetry; Blood Gas Analysis; Liver Disease; Hyperbilirubinemia
MeSH Terms: conditions — Liver Diseases; Hyperbilirubinemia | interventions — Blood Gas Analysis; Oximetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Bilirubin Group (Active Comparator): Low Bilirubin Group: subjects with a bilirubin level less than or equal to 10 mg/dl
  Interventions: Procedure: Arterial Blood Gas; Procedure: Pulse Oximetry Machine; Procedure: Direct and Indirect Serum Bilirubin Measurement
- Medium Bilirubin Group (Active Comparator): Medium Bilirubin Group: subjects with a bilirubin level from 11mg/dl to 30 mg/dl
  Interventions: Procedure: Arterial Blood Gas; Procedure: Pulse Oximetry Machine; Procedure: Direct and Indirect Serum Bilirubin Measurement
- High Bilirubin Group (Active Comparator): High Bilirubin Group: subjects with a bilirubin level greater than or equal to 30 mg/dl
  Interventions: Procedure: Arterial Blood Gas; Procedure: Pulse Oximetry Machine; Procedure: Direct and Indirect Serum Bilirubin Measurement

INTERVENTIONS:
Procedure: Arterial Blood Gas — One blood gas sample will be obtained from an artery in the arm.
  Other Names: ABG
Procedure: Pulse Oximetry Machine — A pulse oximetry machine will be used at one time point to obtain an oxygen saturation reading. This is done by placing a clip onto the finger. The pulse oximetry value displays on the pulse oximeter machine within seconds.
  Other Names: Pulse Ox
Procedure: Direct and Indirect Serum Bilirubin Measurement — One tube of blood will be drawn from a vein in the arm at one timepoint to measure the direct and indirect serum bilirubin levels.
  Other Names: hepatic function panel

SUMMARY:
The purpose of this study is to determine if higher levels of bilirubin in the blood of people with liver disease affects how accurate a pulse oximeter machine is able to measure the concentration of oxygen in the blood. Previous studies have reported conflicting results regarding the affect of high levels of bilirubin in the blood on the accuracy of the pulse oximeter reading. Initial studies showed an underestimation of the oxygen concentration in the presence of elevated bilirubin. Subsequent studies have suggested that high levels of bilirubin in the blood do not influence the accuracy of the pulse oximeter machine. However, recent reports in bone marrow transplant literature and our personal observations in patients with liver disease suggest that high bilirubin levels are associated with an overestimation of the oxygen concentration as measured by the pulse oximeter machine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established liver disease or dysfunction, as determined by abnormal liver function tests, imaging, or biopsy

Exclusion Criteria:

* Patients with unconjugated hyperbilirubinemia, which could be associated with elevations in carboxyhemoglobin
* Patients with poor peripheral perfusion that would compromise accurate pulse oximetric determination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Comparison of pulse oximetric saturation and calculated oxygen saturation. | Enrollment visit

CONTACTS AND LOCATIONS:
Overall Officials: Ram Subramanian, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Staudinger T, Locker GJ, Frass M, Kalhs P. Misleading high values of oxygen saturation measured by pulse oximetry in excessive hyperbilirubinaemia after BMT. Bone Marrow Transplant. 1996 Nov;18(5):1025. No abstract available. PMID 8932862
- [Background] Veyckemans F, Baele P, Guillaume JE, Willems E, Robert A, Clerbaux T. Hyperbilirubinemia does not interfere with hemoglobin saturation measured by pulse oximetry. Anesthesiology. 1989 Jan;70(1):118-22. doi: 10.1097/00000542-198901000-00022. PMID 2912292
- [Background] Ramanathan R, Durand M, Larrazabal C. Pulse oximetry in very low birth weight infants with acute and chronic lung disease. Pediatrics. 1987 Apr;79(4):612-7. PMID 2434913
- [Background] Praud JP, Carofilis A, Bridey F, Lacaille F, Dehan M, Gaultier CL. Accuracy of two wavelength pulse oximetry in neonates and infants. Pediatr Pulmonol. 1989;6(3):180-2. doi: 10.1002/ppul.1950060310. PMID 2470014
- [Background] Ralston AC, Webb RK, Runciman WB. Potential errors in pulse oximetry. III: Effects of interferences, dyes, dyshaemoglobins and other pigments. Anaesthesia. 1991 Apr;46(4):291-5. doi: 10.1111/j.1365-2044.1991.tb11501.x. PMID 2024749
- [Background] Amazon K, Soloni F, Rywlin AM. Separation of bilirubin from hemoglobin by recording derivative spectrophotometry. Am J Clin Pathol. 1981 Apr;75(4):519-23. doi: 10.1093/ajcp/75.4.519. PMID 7223716